CLINICAL TRIAL: NCT04191265
Title: Cardiotoxicity of Aluminum Phosphide Poisoning; Biochemical and Electrophysiological Studies and the Utility of Tropinin and CKmb as Early Biomarkers
Brief Title: Cardiotoxicity of Aluminum Phosphide Poisoning; Tropinin and CKmb as Early Biomarkers
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa Mohamed Abd El-Rahman, Assiut University, Assiut University
Other Study IDs: cardiotoxicity of ALP cases
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Cardiotoxicity; Aluminum Phosphid Poisoning
Keywords: tropinin; CKmb; cardiotoxicity
MeSH Terms: conditions — Cardiotoxicity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: serum tropinin, serum CKmb — early detection of myocardial injury, allowing application of acute cardiac shock and cardiogenic shock

SUMMARY:
Aluminum phosphide (AlP) or rice tablet is a cheap pesticide. When it comes in contact with acid (gastric acid) or moisture, it releases phosphine (PH3) gas. The heart,lungs, liver are the main targets in acute Aluminum phosphide (AlP) poisoning. Most deaths occur due to cardiovascular toxicity.

DETAILED DESCRIPTION:
Aluminium phosphide is a potent respiratory chain enzyme inhibitor. Its most important effect is the inhibition of cytochrome c oxidase. The inhibition of cytochrome c oxidase and other enzymes leads to the generation of superoxide radicals and cellular peroxides , and subsequent cellular injury through lipid peroxidation and other oxidant mechanisms. It stimulates the production of hydrogen peroxide and reactive oxygen species, malonyldialdehyde (MAD), increases superoxide dismutase and inhibits catalase, peroxidase and glutathione . Oxidative stress is one of the main mechanisms of action of aluminium phosphide toxicity

ELIGIBILITY:
Inclusion Criteria: ALP poisoned cases

* admitted with free ECG

Exclusion Criteria:

concomitant ingesion of other drugs or toxins

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Assiut governorate
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2020-06-05 (Estimated); Study Completion 2020-06-05 (Estimated)

PRIMARY OUTCOMES:
assess serum tropinin and CKmb as biomarkers for early detection of ALP induced myocardial injury | 6 months
  assess serum tropinin and CKmb as biomarkers for early detection of ALP induced myocardial injury

CONTACTS AND LOCATIONS:
Locations (1):
- Doaa, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No